CLINICAL TRIAL: NCT04159311
Title: Impact of Osteopathy on IBS-like Symptoms Associated With Ulcerative Colitis in Patients in Remission
Brief Title: Osteopathy on IBS Symptoms in Patients With Ulcerative Colitis in Remission
Acronym: OSTEOMIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study encountered difficulties in including patients
Sponsor: Clinique Paris-Bercy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CParisBercy
Record Dates: First submitted 2019-10-17; First posted 2019-11-12 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Irritable Bowel Syndrome; Ulcerative Colitis
MeSH Terms: conditions — Irritable Bowel Syndrome; Colitis, Ulcerative | interventions — Osteopathic Physicians

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated group (Active Comparator): The "treated group" will have 3 sessions of osteopathy testing followed by osteopathy treatment (M0, M1, M2) and a final testing session at M3.
  Interventions: Other: Osteopathy
- Untreated group (Sham Comparator): The "untreated group" will have 4 sessions of only testing osteopathy (M0, M1, M2, M3).
  Interventions: Other: Osteopathy

INTERVENTIONS:
Other: Osteopathy — testing osteopathy Vs Treating osteopathy

SUMMARY:
Type : interventional, randomized single blind study Aim : to evaluate 3 sessions of osteopathy on IBS-like symptoms associated with ulcerative colitis in remission Number of patients : 50 (randomization 1:1) Duration of the inclusion period : 2 years Primary end-point : Irritable Bowel Syndrome Severity Scoring System (IBS SSS) at 3 months

DETAILED DESCRIPTION:
Osteopathy has been shown to be effective in IBS patients in few studies and to improve IBS-like symptoms in a short series of Crohn patients. IBS-like symptoms are frequent in patients with ulcerative colitis in remission (about 20 %).

The aim of this interventional, randomized single blind study is to evaluate the impact of 3 sessions of osteopathy on Irritable Bowel Syndrome symptoms in 50 patients (randomisation 1:1) with ulcerative colitis in remission (defined by fecal calprotectin < 200 µg/g).

The two group of patients will have 4 sessions of osteopathy (M0, M1, M2, M3). The "treated group" will have 3 sessions of osteopathy testing followed by osteopathy treatment (M0, M1, M2) and a final testing session at M3. The "untreated group" will have 4 sessions of only testing osteopathy (M0, M1, M2, M3).

Primary end-points : Irritable Bowel Syndrome Severity Scoring System (IBS SSS) at 3 months (M3) Secondary end-points : Inflammatory Bowel Disease Questionnaire ol, Functional Assessment of Chronic Illness Therapy-Fatigue at M3, evaluation of osteopathic dysfunctions between M0 and M3, questionnaire for use of medication for IBS between M0 and M3

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 18 and 90
* Patient with ulcerative colitis (whatever the Montreal grade, E1, E2 or E3) In clinical remission for at least 3 months and with fecal calprotectin < 200 µg/g
* No modification of Ulcerative Colitis treatment for at least 3 months
* Patient with IBS-liked symptoms defined as in Rome IV classification for Irritable Bowel Syndrome
* Patient with Irritable Bowel Syndrome Severity Scoring System > 75 at screening
* Patient affiliated to the French Social Security regimen

Exclusion Criteria:

* Patient refusal
* Patient < 18 yoa
* Patient with colonic or ileal stenosis
* Patient diagnosed as undetermined colitis
* Patient not in remission for Ulcerative Colitis as defined by an endoscopic Mayo score > 1 within the 3 months preceding the inclusion and/or fecal calprotectin > 200 µg/g at inclusion
* Osteopathy session(s) within 1 month before inclusion
* Patient with Inflammatory rheumatic disorders (ankylosing spondylitis, psoriatic arthritis, rheumatoid arthritis)
* Patient with Irritable Bowel Syndrome Severity Scoring System <75 at screening
* Patient above 18 yoa with law guardianship

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the score change of Irritable Bowel Syndrome Severity Scoring System (IBS SSS) | Month 1, Month 2, Month 3, Month 4
  index of severity of Irritable Bowel Syndrome symptoms

SECONDARY OUTCOMES:
IBDQol : Inflammatory Bowel Disease Questionnaire | Month 1, Month 2, Month 3, Month 4
  Index of quality of life dedicated to Inflammatory Disease Bowel patients : the score is high, better the quality of life
FACIT-F : Functional Assessment of Chronic Illness Therapy-Fatigue | Month 1, Month 2, Month 3, Month 4
  Validated fatigue score with question about quality of life 45/5000
  if the score is high, the patient is tired
Evaluation of osteopathic dysfunctions | Month 1, Month 2, Month 3, Month 4
  it will be interesting to see if patients with remission-prone RCH have similar osteopathic dysfunctions at the beginning of the study, and then if the management during the study influences or not these osteopathic dysfunctions.
  Osteopathic dysfunction is an alteration of the mobility, viscoelasticity or texture of somatic system components. It is accompanied or not by a painful sensibility.
Questionnaire for use of medication for Irritable Bowel Syndrome | Month 1, Month 2, Month 3, Month 4
  if treatment modification, dose reduction or change in treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maryan Cavicchi, MD, PhD, Study Director — Clinique Paris-Bercy
Locations (1):
- Clinique Paris Bercy, Charenton-le-Pont, France

IPD SHARING:
Plan to Share IPD: No